CLINICAL TRIAL: NCT00531843
Title: The Use of Fondaparinux in Preventing Thromboembolism in High Risk Trauma Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mary Knudson, M.D. (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Mary Knudson, M.D., Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H6693-30799-01
Record Dates: First submitted 2007-09-17; First posted 2007-09-19 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-10

CONDITIONS: Venous Thromboembolism
Keywords: deep vein thrombosis; venous thromboembolism; pulmonary embolism
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1A (Experimental): Patients at high risk for venous thromboembolism (criteria: age>=40, pelvic fracture, lower extremity fracture, shock on presentation, spinal cord injury, head injury with Abbreviated Injury Scale (AIS) >=3). These patients will receive fondaparinux 2.5mg via subcutaneous administration (SubQ) daily.
  Interventions: Drug: fondaparinux sodium
- 1B (Active Comparator): Patients at high risk for venous thromboembolism (criteria: age>=40, pelvic fracture, lower extremity fracture, shock on presentation, spinal cord injury, head injury with AIS >=3) who also have a contraindication to anticoagulant(enoxaparin)administration such as renal failure with creatine clearance <30 mL/min, head injury with head AIS >=3), uncontrolled hemorrhage, uncorrected coagulopathy, persistent thrombocytopenia. These patients will receive mechanical compression.
  Interventions: Device: sequential compression devices
- 2A (Experimental): Patients at very high risk for venous thromboembolism (criteria: major operative procedure, venous injury, ventilator days >3, 2 or more high risk factors). These patients will receive fondaparinux 2.5mg SubQ daily and mechanical compression.
  Interventions: Drug: fondaparinux sodium
- 2B (Active Comparator): Patients at very high risk for venous thromboembolism (criteria: major operative procedure, venous injury, ventilator days >3, 2 or more high risk factors) who also have a contraindication to anticoagulant(enoxaparin)administration such as renal failure creatine clearance <30 mL/min, head injury with head AIS >=3), uncontrolled hemorrhage, uncorrected coagulopathy, persistent thrombocytopenia. These patients will receive mechanical compression and possibly temporary inferior vena cava (IVC) filter(as determined by the patient's care givers).
  Interventions: Device: sequential compression devices

INTERVENTIONS:
Drug: fondaparinux sodium — fondaparinux 2.5mg SubQ daily for DVT prophylaxis to be started by treating physicians once deemed safe and to be discontinued once patient in discharged from the hospital or at discretion of treating physicians.
  Other Names: Arixtra
  Arms: 1A; 2A
Device: sequential compression devices — Sequential compression devices at all times during the patient's hospital admission will be used in patients who have a contraindication to pharmacologic DVT prophylaxis. This is already the current standard of care.
  Other Names: Arixtra
  Arms: 1B; 2B

SUMMARY:
Trauma patients are at high risk of developing deep vein thrombosis (DVT) and pulmonary embolism (PE). The incidence of DVT varies greatly from 5-63% among studies depending on patient's individual risk factors, modality of prophylaxis, and methods of detection. The incidence of PE may be as low (0.3-4.3%) but carries a mortality of 20-50% which makes prevention of DVT of the utmost importance. The current standard of care for DVT prophylaxis in the trauma patient with high risk of DVT is enoxaparin, a low molecular weight heparin, administered twice a day as long as anticoagulation in not contraindicated. Many studies have demonstrated its efficacy when compared to mechanical compression and to unfractionated heparin, however one of the most robust of these studies still reported an DVT incidence of 35% in patients treated with enoxaparin. Another drug, fondaparinux, is a selective factor Xa inhibitor that could offer added benefits over enoxaparin such as once daily dosing and a drastically reduced risk of heparin induced thrombocytopenia (HIT). Fondaparinux has been already be widely used in post-operative hip surgery and major knee surgery patients with good results. It has also been shown to be effective in DVT prophylaxis in patients who have had major abdominal surgery and also in acute medical patients. Fondaparinux has yet to be used in trauma patients. Trauma patients are a diverse and distinct population given the acuity of their injuries and their increased risk of bleeding who at this time still do not have a perfect method for DVT prophylaxis. We hypothesize that fondaparinux will be effective in decreasing the risk of DVT when used in the trauma patient population. This is a non randomized prospective cohort study designed to test the efficacy of fondaparinux in the prophylaxis of DVT and PE in trauma patients.

DETAILED DESCRIPTION:
Patients with trauma admitted to San Francisco General Hospital and qualify for the study will be assigned to +fondaparinux and no fondaparinux arms based on guidelines that were developed for and are considered the standard of care for the use of low molecular weight heparin in the same group of patients for the same indication. These guidelines will separate patients at risk for DVT into those that are high risk and very high risk. The primary efficacy outcome measures will be DVT and PE. Presence of DVT will be assessed with serial color flow duplex ultrasound during the patients in hospital stay at weekly intervals up to 3 weeks and when the patient has symptoms of DVT. PE will be diagnosed according to clinical suspicion by the patients treating physicians and subsequent imaging by CT. We plan on enrolling approximately 100 patients in the +fondaparinux and 100 patients in the no fondaparinux arm. We will compare both the incidence of DVT and PE in these groups and to the incidences in the literature and historical controls. A second aim of the study is to evaluate the adverse outcomes such as increased bleeding in patients who receive fondaparinux. A third and final aim of the study is to describe the effect of fondaparinux on antifactor Xa levels in trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18 years old admitted to San Francisco General Hospital for injury with at least one risk factor for venous thromboembolism (VTE).

Risk factors are: Age ≥ 40 years, pelvic fracture, lower extremity fracture, spinal cord injury, shock or head injury, major operative procedure, mechanical ventilation > 3 days, venous injury

Exclusion Criteria:

* prisoners
* pregnant patients
* patients who are anticipated to have a < 5 day length of stay as determined by the admitting trauma surgeon
* patients who decline to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Margaret Knudson, MD, Principal Investigator — The University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Agnelli G, Bergqvist D, Cohen AT, Gallus AS, Gent M; PEGASUS investigators. Randomized clinical trial of postoperative fondaparinux versus perioperative dalteparin for prevention of venous thromboembolism in high-risk abdominal surgery. Br J Surg. 2005 Oct;92(10):1212-20. doi: 10.1002/bjs.5154. PMID 16175516
- [Background] Geerts WH, Jay RM, Code KI, Chen E, Szalai JP, Saibil EA, Hamilton PA. A comparison of low-dose heparin with low-molecular-weight heparin as prophylaxis against venous thromboembolism after major trauma. N Engl J Med. 1996 Sep 5;335(10):701-7. doi: 10.1056/NEJM199609053351003. PMID 8703169
- [Background] Velmahos GC. Posttraumatic thromboprophylaxis revisited: an argument against the current methods of DVT and PE prophylaxis after injury. World J Surg. 2006 Apr;30(4):483-7. doi: 10.1007/s00268-005-0427-9. PMID 16568226
- [Background] Hill AB, Garber B, Dervin G, Howard A. Heparin prophylaxis for deep venous thrombosis in a patient with multiple injuries: an evidence-based approach to a clinical problem. Can J Surg. 2002 Aug;45(4):282-7. PMID 12174986
- [Background] Geerts WH, Pineo GF, Heit JA, Bergqvist D, Lassen MR, Colwell CW, Ray JG. Prevention of venous thromboembolism: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):338S-400S. doi: 10.1378/chest.126.3_suppl.338S. PMID 15383478
- [Background] Turpie AG, Bauer KA, Eriksson BI, Lassen MR; PENTATHALON 2000 Study Steering Committee. Postoperative fondaparinux versus postoperative enoxaparin for prevention of venous thromboembolism after elective hip-replacement surgery: a randomised double-blind trial. Lancet. 2002 May 18;359(9319):1721-6. doi: 10.1016/S0140-6736(02)08648-8. PMID 12049860
- [Background] Kudsk KA, Fabian TC, Baum S, Gold RE, Mangiante E, Voeller G. Silent deep vein thrombosis in immobilized multiple trauma patients. Am J Surg. 1989 Dec;158(6):515-9. doi: 10.1016/0002-9610(89)90182-7. PMID 2589580
- [Background] Knudson MM, Ikossi DG. Venous thromboembolism after trauma. Curr Opin Crit Care. 2004 Dec;10(6):539-48. doi: 10.1097/01.ccx.0000144941.09650.9f. PMID 15616398
- [Background] Donat F, Duret JP, Santoni A, Cariou R, Necciari J, Magnani H, de Greef R. The pharmacokinetics of fondaparinux sodium in healthy volunteers. Clin Pharmacokinet. 2002;41 Suppl 2:1-9. doi: 10.2165/00003088-200241002-00001. PMID 12383039
- [Background] Knudson MM, Ikossi DG, Khaw L, Morabito D, Speetzen LS. Thromboembolism after trauma: an analysis of 1602 episodes from the American College of Surgeons National Trauma Data Bank. Ann Surg. 2004 Sep;240(3):490-6; discussion 496-8. doi: 10.1097/01.sla.0000137138.40116.6c. PMID 15319720
- [Background] Eriksson BI, Bauer KA, Lassen MR, Turpie AG; Steering Committee of the Pentasaccharide in Hip-Fracture Surgery Study. Fondaparinux compared with enoxaparin for the prevention of venous thromboembolism after hip-fracture surgery. N Engl J Med. 2001 Nov 1;345(18):1298-304. doi: 10.1056/NEJMoa011100. PMID 11794148
- [Background] Bauer KA, Eriksson BI, Lassen MR, Turpie AG; Steering Committee of the Pentasaccharide in Major Knee Surgery Study. Fondaparinux compared with enoxaparin for the prevention of venous thromboembolism after elective major knee surgery. N Engl J Med. 2001 Nov 1;345(18):1305-10. doi: 10.1056/NEJMoa011099. PMID 11794149
- [Background] Geerts WH, Code KI, Jay RM, Chen E, Szalai JP. A prospective study of venous thromboembolism after major trauma. N Engl J Med. 1994 Dec 15;331(24):1601-6. doi: 10.1056/NEJM199412153312401. PMID 7969340
- [Background] Allen TL, Carter JL, Morris BJ, Harker CP, Stevens MH. Retrievable vena cava filters in trauma patients for high-risk prophylaxis and prevention of pulmonary embolism. Am J Surg. 2005 Jun;189(6):656-61. doi: 10.1016/j.amjsurg.2005.03.003. PMID 15910715
- [Background] Cohen AT, Davidson BL, Gallus AS, Lassen MR, Prins MH, Tomkowski W, Turpie AG, Egberts JF, Lensing AW; ARTEMIS Investigators. Efficacy and safety of fondaparinux for the prevention of venous thromboembolism in older acute medical patients: randomised placebo controlled trial. BMJ. 2006 Feb 11;332(7537):325-9. doi: 10.1136/bmj.38733.466748.7C. Epub 2006 Jan 26. PMID 16439370
- [Result] Lu JP, Knudson MM, Bir N, Kallet R, Atkinson K. Fondaparinux for prevention of venous thromboembolism in high-risk trauma patients: a pilot study. J Am Coll Surg. 2009 Nov;209(5):589-94. doi: 10.1016/j.jamcollsurg.2009.08.001. Epub 2009 Sep 11. PMID 19854398

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During a 6-month period, consecutive adults presenting to one Level I urban trauma center were screened for eligibility, enrolled and assigned to a treatment category using previously-developed clinical guidelines.
Pre-assignment Details: Of 105 enrolled participants, 18 were excluded from analysis (13 discharged or transferred prior to second venous ultrasonography; 4 received non-study DVT prophylaxis; 1 had a known protein-C deficiency).
Groups:
- Fondaparinux Sodium: Patients at high risk or very high risk for venous thromboembolism received fondaparinux 2.5mg via subcutaneous administration (SubQ) daily, with (very high risk) or without (high risk) mechanical compression upon admission or by 3rd day after injury.
- No Fondaparinux: Patients at high risk or very high risk for venous thromboembolism AND contraindication to anticoagulant administration received mechanical compression, with (very high risk) or without (high risk) possible temporary inferior vena cava (IVC) filter (prn as determined by caregiver).
Period: Overall Study
Arm/Group | Fondaparinux Sodium | No Fondaparinux
Started | 81 | 6
Completed | 81 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fondaparinux Sodium: Patients at high risk or very high risk for venous thromboembolism received fondaparinux 2.5mg SubQ daily, with (very high risk) or without (high risk) mechanical compression upon admission or by 3rd day after injury.
- No Fondaparinux: Patients at high risk or very high risk for venous thromboembolism AND contraindication to anticoagulant administration received mechanical compression, with (very high risk) or without (high risk) possible temporary IVC filter (prn as determined by caregiver).
- Total: Total of all reporting groups
Arm/Group | Fondaparinux Sodium | No Fondaparinux | Total
Number analyzed (Participants) | 81 | 6 | 87
Age Continuous [Mean (Standard Deviation); unit: years] | 43.1 (19.3) | 56.8 (20.9) | 44.3 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 1 | 22
  Male | 60 | 5 | 65
Region of Enrollment [Number; unit: participants]
  United States | 81 | 6 | 87

OUTCOME MEASURES:

1. Secondary Outcome: Normal Trough and Peak Fondaparinux Concentration
Description: Serum samples were collected 30 minutes before (trough) and 2 hours after (peak) the third dose of fondaparinux. Normative data plots comparing study participants with healthy volunteers were supplied by the company outsourced to analyze samples.
Time Frame: Day 3
Population: Serum samples were obtained from 63 representative patients from our study who received Fondaparinux and compared against normative values from normal volunteers supplied by our sponsor.
Measure: Number; unit: Participants
Arm/Group | Fondaparinux Sodium | No Fondaparinux
Number analyzed (Participants) | 63 | 0
Participants
  Trough values outside normative range | 0 |
  Peak values outside normative range | 0 |

2. Primary Outcome: Presence of Deep Vein Thrombosis (DVT) or Pulmonary Embolus (PE)
Description: Color-flow duplex venous ultrasonography examinations of upper and lower extremities were performed within 48 hours of injury, and then weekly until discharge or 3 weeks. DVT was defined as any clot occurring in the subclavian, iliac, femoral, or popliteal location. Patients were examined daily for clinical signs and symptoms of venous thromboembolism (VTE) and PE. Small, nonocclusive clots discovered in other locations were observed for progression on sequential ultrasonography examinations.
Time Frame: within 3 weeks post injury
Population: Of 11 patients with initial contraindication to anticoagulation, 5 were cleared by the treating physicians to receive fondaparinux within 3 days of injury, and 6 were not.
Measure: Number; unit: participants
Arm/Group | Fondaparinux Sodium | No Fondaparinux
Number analyzed (Participants) | 81 | 6
participants
  DVT | 2 | 2
  DVT after fondaparinux | 1 | NA — This arm/group did not receive Fondaparinux.
  PE | 0 | 0

3. Secondary Outcome: Increased Bleeding Attributed to Fondaparinux
Description: Coagulopathic bleeding due to fondaparinux was suspected in patients requiring packed red cell transfusions after initiation of fondaparinux therapy only if the change in hematocrit prompting transfusion was not clinically commensurate with the degree of injuries that the patient had sustained (primarily orthopaedic) and/or the hematocrit did not respond appropriately post-transfusion.
Time Frame: 3 weeks post injury
Measure: Number; unit: participants
Arm/Group | Fondaparinux Sodium | No Fondaparinux
Number analyzed (Participants) | 81 | 0
participants | 0 |

ADVERSE EVENTS:
Time Frame: 3 weeks post-injury
Description: This study did not record adverse events that were related to the severity of participants' trauma unless assessed for potential attribution to study participation
Arm/Group | Fondaparinux Sodium | No Fondaparinux
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/6
Other Adverse Events (participants affected / at risk) | 13/81 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fondaparinux Sodium (N=81) | No Fondaparinux (N=6)
Drop in hematocrit (Blood and lymphatic system disorders) | 13 (13) | 0 (0)
DVT (Vascular disorders) | 2 (2) | 2 (2)
Superficial nonoccluding clots (Vascular disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes